CLINICAL TRIAL: NCT01857258
Title: Green Tea Confections For Managing Postprandial Hyperglycemia-Induced Vascular Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013H0116
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Hyperglycemia; Cardiovascular Disease
Keywords: green tea; catechins; vascular endothelial function; postprandial hyperglycemia; oxidative stress
MeSH Terms: conditions — Hyperglycemia; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green Tea (Experimental): Participants will be provided a confection containing green tea concentrate
  Interventions: Dietary Supplement: Green Tea Concentrate
- Control (Active Comparator): Participants will be provided a confection devoid of green tea concentrate
  Interventions: Dietary Supplement: Green Tea Concentrate

INTERVENTIONS:
Dietary Supplement: Green Tea Concentrate — Green tea concentrate is being examined as a dietary supplement that can regulate postprandial excursions in blood glucose

SUMMARY:
The objective of this study is to formulate and validate a green tea confection (i.e. "gummy" candy) as a strategy to attenuate postprandial hyperglycemia-induced impairments in vascular function. The central hypothesis is that a green tea confection will protect against vascular endothelial dysfunction by suppressing postprandial hyperglycemia. The central hypothesis of this application will be assessed by developing a green tea-containing confection, examining its physiochemical properties and its inhibition of starch digestion, and then validating its vasoprotective activities in healthy humans by assessing its blood glucose-regulating activities.

DETAILED DESCRIPTION:
The study involves validating a green tea confection (i.e. "gummy" candy) as a dietary strategy to attenuate postprandial hyperglycemia-induced impairments in vascular function. The central hypothesis is that a green tea confection will protect against vascular endothelial dysfunction by suppressing postprandial hyperglycemia. The central hypothesis of this application will be assessed by providing research participants 75 grams of carbohydrate in the form of a confection that contains no green tea concentrate or green tea concentrate at a level equivalent to approximately 3 cups of freshly brewed tea. Blood glucose and brachial artery flow-mediated dilation will be assessed at regular intervals during the 3 hour postprandial period to define the extent to which green tea attenuates postprandial increases in blood glucose and decreases in vascular function that otherwise occur in a hyperglycemia-dependent manner.

ELIGIBILITY:
Inclusion Criteria:

* Plasma glucose <100 mg/dL
* Plasma total cholesterol <200 mg/dL
* Plasma triglycerides <140 mg/dL
* Blood pressure <140/90
* non-dietary supplement user for >2 months
* no use of medications known to affect carbohydrate metabolism,
* nonsmoker / never smoker
* no history of cardiovascular disease or gastrointestinal disorders

Exclusion Criteria:

* allergies or aversions to green tea and/or corn starch,
* excessive alcohol consumption (>3 drinks/d),
* >5 h/wk of aerobic activity

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sapper TN, Mah E, Ahn-Jarvis J, McDonald JD, Chitchumroonchokchai C, Reverri EJ, Vodovotz Y, Bruno RS. A green tea-containing starch confection increases plasma catechins without protecting against postprandial impairments in vascular function in normoglycemic adults. Food Funct. 2016 Sep 14;7(9):3843-53. doi: 10.1039/c6fo00639f. Epub 2016 Aug 5. PMID 27494176

RESULTS

PARTICIPANT FLOW:
Groups:
- Green Tea First, Then Control: Participants will be provided a confection containing green tea concentrate in fasting state one time. After a washout period of 7 days, they then will be provided a confection devoid of green tea concentrate in fasting state one time.
  The green tea concentrate is being examined as a dietary supplement that can regulate postprandial excursions in blood glucose. The confection provides 50 grams of starch and 1 gram of green tea concentrate.
- Control First, Then Green Tea: Participants will be provided a confection devoid of green tea concentrate in fasting state one time. After a washout period of 7 days, they then will be provided a confection containing green tea concentrate in fasting state one time.
  The green tea concentrate is being examined as a dietary supplement that can regulate postprandial excursions in blood glucose. The confection provides 50 grams of starch and 1 gram of green tea concentrate.
Period: First Intervention (3 h Postprandially)
Arm/Group | Green Tea First, Then Control | Control First, Then Green Tea
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Wash-out Period (7 Days)
Arm/Group | Green Tea First, Then Control | Control First, Then Green Tea
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention (3 h Postprandially)
Arm/Group | Green Tea First, Then Control | Control First, Then Green Tea
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Participant Characteristics: All participants completed both arms of the cross-over study
Arm/Group | Baseline Participant Characteristics
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.4 (1.8)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 88.9 (5.2)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 160.5 (21.44)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Blood Glucose
Description: Blood glucose will be measured at 0, 30, 60, 90, 120, 150 and 180 minutes following the ingestion of a confection to calculate area under the concentration-time curve.
Time Frame: Area under the Curve, 0, 30, 60, 90, 120, 150, 180 minutes post-dose
Measure: Mean (Standard Error); unit: mmol/L * min
Arm/Group | Green Tea | Control
Number analyzed (Participants) | 15 | 15
mmol/L * min | 998 (29) | 981 (28)

2. Primary Outcome: Area Under the Curve of Brachial Artery Flow Mediated Dilatiion
Description: Brachial artery flow-mediated dilation will be measured at 0, 30, 60, 90, 120, 150, and 180 minutes following the ingestion of a confection.
Time Frame: Area under the Curve, 0, 30, 60, 90, 120, 150, 180 minutes post-dose
Measure: Mean (Standard Error); unit: %FMD * min
Arm/Group | Green Tea | Control
Number analyzed (Participants) | 15 | 15
%FMD * min | 614 (65) | 653 (66)

3. Primary Outcome: Brachial Artery Flow-mediated Dilation
Time Frame: 0 min (baseline)
Measure: Mean (Standard Error); unit: % dilation
Arm/Group | Control | Green Tea
Number analyzed (Participants) | 15 | 15
% dilation | 3.71 (0.42) | 3.54 (0.42)

4. Primary Outcome: Brachial Artery Flow-mediated Dilation
Time Frame: 60 min
Measure: Mean (Standard Error); unit: % dilation
Arm/Group | Control | Green Tea
Number analyzed (Participants) | 15 | 15
% dilation | 3.23 (0.44) | 3.04 (0.35)

5. Secondary Outcome: Malondialdehyde (0 Min)
Time Frame: Baseline (0 min)
Measure: Mean (Standard Error); unit: uM
Arm/Group | Green Tea | Control
Number analyzed (Participants) | 15 | 15
uM | 1.18 (0.15) | 1.18 (0.16)

6. Secondary Outcome: Malondialdehyde
Time Frame: 60 min postprandially
Measure: Mean (Standard Error); unit: uM
Arm/Group | Green Tea | Control
Number analyzed (Participants) | 15 | 15
uM | 1.44 (0.15) | 1.47 (0.14)

7. Secondary Outcome: Ratio of Asymmetric Dimethylarginine Relative to Arginine
Time Frame: 0 min (baseline)
Measure: Mean (Standard Error); unit: nmol/umol
Arm/Group | Control | Green Tea
Number analyzed (Participants) | 15 | 15
nmol/umol | 5.75 (0.26) | 6.24 (0.42)

8. Secondary Outcome: Ratio of Asymmetric Dimethylarginine Relative to Arginine
Time Frame: 60 min (baseline)
Measure: Mean (Standard Error); unit: nmol/umol
Arm/Group | Control | Green Tea
Number analyzed (Participants) | 15 | 15
nmol/umol | 6.96 (0.51) | 7.18 (0.53)

ADVERSE EVENTS:
Time Frame: Participants were monitored for any adverse events in response to ingesting starch-based confections containing no green tea or with green tea through study completion (9 days).
Groups:
- Green Tea, Then Control: Participants will be provided a confection containing green tea concentrate in fasting state one time. After a washout period of 7 days, they then will be provided a confection devoid of green tea concentrate in fasting state one time.
  Green Tea Concentrate: Green tea concentrate is being examined as a dietary supplement that can regulate postprandial excursions in blood glucose
- Control, Then Green Tea: Participants will be provided a confection devoid of green tea concentrate in fasting state one time. After a washout period of 7 days, they then will be provided a confection containing green tea concentrate in fasting state one time.
  Green Tea Concentrate: Green tea concentrate is being examined as a dietary supplement that can regulate postprandial excursions in blood glucose
Arm/Group | Green Tea, Then Control | Control, Then Green Tea
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
This study was limited to normoglycemic adults who were healthy. Future studies may consider populations having glucose intolerance to examine the extent to which green tea attenuates starch-induced hyperglycemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No